CLINICAL TRIAL: NCT00929721
Title: Global Active Surveillance for Community-Acquired Pneumonia (CAP) in Adults 50 Years and Older
Brief Title: A Global Active Surveillance for Community Acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 6115A1-4000
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Community Acquired Pneumonia
Keywords: CAP
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Blood Specimen Collection; X-Rays; Urine Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with Community-Acquired Pneumonia (Other): Subjects with Community-Acquired Pneumonia
  Interventions: Procedure: Blood draw; Procedure: Chest X-ray; Procedure: urine specimen; Procedure: Nasopharyngeal swab; Procedure: sputum

INTERVENTIONS:
Procedure: Blood draw — culture for Streptococcus pneumoniae Frequency-1
  Other Names: Blood stick
Procedure: Chest X-ray — image of the lungs to assess changes consistent with pneumonia Frequency-1
  Other Names: Picture of lungs
Procedure: urine specimen — assay for the presence of Streptococcus pneumoniae Binax and UAD
  Other Names: urine dipstick test
Procedure: Nasopharyngeal swab — culture for Streptococcus pneumoniae Frequency-1
  Other Names: swab from inside the nose and throat
Procedure: sputum — culture for Streptococcus pneumoniae Frequency-1
  Other Names: collection secretions produced during cough

SUMMARY:
This study is an observational surveillance study to identify adults 50 years and older who present to a study healthcare facility with signs and symptoms of Community-Acquired Pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 50 years of age or older
* Subject must reside in the surveillance area
* Subjects who present to a study healthcare facility where the treating physician clinically suspects CAP

Exclusion Criteria:

* Any subject who is transferred to a study healthcare facility after already being hospitalized for 48 hours or more at any other in-patient facility (such as a community hospital).
* Hospital Acquired pneumonia (ie, develops signs and symptoms of pneumonia after being hospitalized for 48 hours or more).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5172 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence rates of CAP in adults 50 years and older | up to 120 days from enrollment

SECONDARY OUTCOMES:
Frequency of bacterial agents associated with CAP, Case fatality and incidence rates of CAP number and characteristics of subjects from outpatient clinics, emergency rooms, and hospital in-patient departments | up to 120 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Chrzanów, Poland

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-4000&StudyName=A%20Global%20Active%20Surveillance%20for%20Community%20Acquired%20Pneumonia